CLINICAL TRIAL: NCT00745940
Title: A Multi-site, Randomized, Controlled Trial of a Mindfulness-based Cognitive Therapy Intervention for Treating Depression in a Traumatic Brain Injury Population.
Brief Title: Mindfulness-Based Cognitive Therapy Intervention to Treat Depression in Individuals With a Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lakehead University (Other)
Collaborators: Ontario Neurotrauma Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ABI-MIND2-476
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Results first posted 2014-02-17 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-02

CONDITIONS: Depression; Traumatic Brain Injury
Keywords: Mindfulness-Based Cognitive Therapy; MBCT; Depression; Traumatic Brain Injury; TBI
MeSH Terms: conditions — Depression; Brain Injuries, Traumatic | interventions — Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MBCT Intervention Group (Experimental): The curriculum of our mindfulness intervention draws upon elements from the mindfulness-based stress reduction program, and Segal and colleagues manual for mindfulness-based cognitive therapy. It was modified by one of the investigators to address issues associated with traumatic brain injury (e.g., problems with attention, concentration, memory, fatigue). The intervention was increased to ten weeks with one and a half hour weekly sessions, along with a 20-30 minute daily meditation home practice. Further adaptations included simplified language, the use of repetition to reinforce concepts, and visual aids. More attention was paid to fostering learning conditions to encourage an environment of trust and non-judgement. Connections between learning activities was also made more explicit.
  Interventions: Behavioral: MBCT for TBI
- MBCT Control Group (No Intervention): Control group waited.

INTERVENTIONS:
Behavioral: MBCT for TBI — Subjects will participate in a 10-week Mindfulness-Based Cognitive Therapy Program led by two trained facilitators. Weekly one-and-a-half hour group sessions will guide subjects through exercises such as meditation, awareness, and breathing techniques aimed at developing skills to help with tension, stress, anxiety and depression. Subjects will be encouraged to practice skills at home and in daily life.
  Other Names: MBCT
  Arms: MBCT Intervention Group

SUMMARY:
The purpose of this study is to determine whether mindfulness-based cognitive therapy is effective in reducing depression symptoms in individuals who have experienced a traumatic brain injury.

The investigators hypothesize that participants who are given the ten-week intervention will have fewer depression symptoms than the participants in the control group, and this improvement will be maintained at the three-month follow-up assessment.

DETAILED DESCRIPTION:
Major depression is a significant chronic problem for people with traumatic brain injury (TBI), and its treatment is difficult. A promising approach to treat depression is mindfulness-based cognitive therapy (MBCT), a relatively new therapeutic approach rooted in mindfulness-based stress-reduction (MBSR) and cognitive behavioural therapy (CBT). This multi-site, randomized, controlled trial of a MBCT intervention will examine the value of this intervention in improving quality of life and decreasing depression in people with TBI. MBCT may represent a time-limited, cost-effective group intervention through which clinicians would have an opportunity to address some of the most debilitating aspects of TBI.

ELIGIBILITY:
Inclusion Criteria:

* traumatic brain injury suffered more than one year ago but less than five
* Evidence of depression post-traumatic brain injury (Beck Depression Inventory-II score of 16 or greater)
* Ability to speak and read English
* Age 18 or more

Exclusion Criteria:

* Inability to benefit from the intervention based a consensus process amongst study clinical psychologist and physicians, and from scores on memory and auditory attention (California Verbal Learning Test, Digit Span subsection of Wechsler Adult Intelligence Scale); verbal fluency and executive functioning (Controlled Oral Word Association Test); verbal abstract reasoning (Similarities subsection of Wechsler Adult Intelligence Scale); and executive functioning (Trail Making Test).
* Evidence of unusual psychological processes such as psychosis, suicidal ideation, substance abuse, or major concurrent mental illness (Beck Depression Inventory-II and Symptom Checklist-90-R will supplement the decision-making process of study clinicians).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2009-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Bédard, PhD, Principal Investigator — Lakehead University
Locations (3):
- Canada (3):
  - Ottawa Hospital Rehabilitation Centre, Ottawa, Ontario
  - St. Joseph's Care Group, Thunder Bay, Ontario
  - Toronto Rehabilitation Institute, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were sought from local sources including: outpatient programs/clinics for individuals with neurological injury, newspaper and television advertisements, a brain injury association, social events related to treatment of brain injury, as well as through appeals to family physicians, psychologists, chiropractors and nurse practitioners.
Period: Overall Study
Arm/Group | MBCT Intervention Group | MBCT Control Group
Started | 57 | 48
Completed | 38 | 38
Not Completed | 19 | 10

BASELINE CHARACTERISTICS:
Population: We initially had 57 MBCT Intervention group participants and 48 Control group participants. 29 participants (28%) did not complete the study - 17 prior to their respective arm starting and 8 during the intervention. Thus, for our analysis we had 38 in each arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | MBCT Intervention Group | MBCT Control Group | Total
Number analyzed (Participants) | 38 | 38 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 38 | 76
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.10 (12.03) | 45.81 (14.80) | 46.46 (13.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 15 | 34
  Male | 19 | 23 | 42
Region of Enrollment [Number; unit: participants]
  Canada | 38 | 38 | 76

OUTCOME MEASURES:

1. Secondary Outcome: Patient Health Questionnaire (PHQ-9)
Description: The PHQ-9 is a self-administered questionnaire based on the PRIME-MD diagnostic instrument for common mental disorders. Each of the 9 DSM-IV criteria is scored on a four point Likert scale ranging from "0" (not at all) to "3" (nearly every day) with higher scores indicative of greater depression symptoms. Scores range from a low of 0 to a high of 27.
Time Frame: Baseline data were collected prior to the intervention and post-intervention data were collected 10 weeks later.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MBCT Intervention Group | MBCT Control Group
Number analyzed (Participants) | 38 | 38
units on a scale
  Baseline Score on PHQ-9 (total score) | 11.53 (5.03) | 14.08 (6.52)
  Post Intervention Score on PHQ-9 (total score) | 10.19 (5.88) | 12.84 (6.74)

2. Primary Outcome: Beck Depression Inventory - II
Description: The Beck Depression Inventory (BDI-II) is a 21-question multiple-choice self-report inventory, one of the most widely used instruments for measuring the severity of depression. It assesses the intensity of depression into 4 categories ranging from minimal (scores from 0-13) to severe (scores from 29-63) (79). Each item is a list of four statements arranged in increasing severity about a particular symptom of depression. The depression criteria are consistent with those of the Diagnostic and Statistical Manual of Mental Health Disorders-Fourth Edition (DSM-IV). The cognitive-affective factor includes items concerning sadness, past failure, loss of pleasure, guilty feelings, punishment feelings, self-dislike, self-criticalness, suicidal thoughts or wishes, crying, agitation, loss of interest, worthlessness, and irritability. The somatic factor is comprised of loss of energy, changes in sleeping pattern, changes in appetite, concentration difficulty, and tiredness or fatigue.
Time Frame: Baseline data were collected prior to the intervention and post-intervention data were collected 10 weeks later.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MBCT Intervention Group | MBCT Control Group
Number analyzed (Participants) | 38 | 38
units on a scale
  Baseline Score on BDI-II (total score) | 25.47 (8.12) | 27.13 (10.61)
  Post Intervention Score on the BDI-II (total score | 18.84 (10.26) | 25.00 (13.12)

3. Secondary Outcome: Symptom Checklist-90 Revised (Depression Subscale)
Description: The Symptom Checklist-90 Revised (SCL-90-R) is a 90 item self-report questionnaire designed to measure nine primary symptom dimensions: somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, and psychoticism from the last two weeks from the current point in time. A five point Likert scale is used ranging from "Not at All" to "Extremely" with higher scores indicative of greater symptoms. There are 13 questions in the depression subscale with scores ranging between 0 and 52. To help with interpretation of all SCL-90-R sub-scales, we transformed this sub-scale total score back to a score between 0 to 4 with higher scores indicating greater depression symptoms.
Time Frame: Baseline data were collected prior to the intervention and post-intervention data were collected 10 weeks later.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MBCT Intervention Group | MBCT Control Group
Number analyzed (Participants) | 38 | 38
units on a scale
  Baseline Symptom Checklist-90-R (Depression) | 1.62 (0.80) | 1.36 (0.90)
  Post Intervention Symptom Checkl-90-R (Depression) | 1.74 (0.94) | 1.49 (1.04)

4. Secondary Outcome: Philadelphia Mindfulness Scale (Awareness Subscale)
Description: The Philadelphia Mindfulness Scale (PHLMS) is a measure of mindfulness to assess present-moment awareness and acceptance. The questionnaire comprises 20 questions rated on a five-point Likert scale with higher scores indicative of greater mindfulness. It comprises two subscales - Awareness and Acceptance. The range of scores on the Awareness subscale is 10 to 50 and the range on the Acceptance subscale is 10 to 50 with higher scores indicative a greater awareness and acceptance respectively.
Time Frame: Baseline data were collected prior to the intervention and post-intervention data were collected 10 weeks later.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MBCT Intervention Group | MBCT Control Group
Number analyzed (Participants) | 38 | 38
units on a scale
  Baseline Score on PHLMS (Awareness Subscale) | 33.84 (6.62) | 33.97 (6.02)
  Post Intervention Score on PHLMS (Awareness) | 35.10 (6.01) | 34.42 (5.17)

5. Secondary Outcome: Philadelphia Mindfulness Scale (Acceptance Subscale)
Description: as for outcome 4
Time Frame: Baseline data were collected prior to the intervention and post-intervention data were collected 10 weeks later.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MBCT Intervention Group | MBCT Control Group
Number analyzed (Participants) | 38 | 38
units on a scale
  Baseline Score on PHLMS (Acceptance Subscale) | 28.35 (7.42) | 28.14 (7.45)
  Post Intervention Score on PHLMS (Acceptance) | 31.16 (7.35) | 29.39 (7.55)

ADVERSE EVENTS:
Arm/Group | MBCT Intervention Group | MBCT Control Group
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/48
Other Adverse Events (participants affected / at risk) | 0/57 | 0/48

LIMITATIONS AND CAVEATS:
It is not possible to generalize our findings to the general population of people with a traumatic brain injury. Participants self-selected. Some did not complete the intervention. The control group was a "wait-list" control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No